CLINICAL TRIAL: NCT06223490
Title: Effect of Cryolipolysis on Insulin Resistance in Type 2 Diabetic Females With Abdominal Obesity
Brief Title: Effect of Cryolipolysis on Insulin Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noura Ramadan Fahmy, Resident of Physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Noura Fahmy
Record Dates: First submitted 2024-01-06; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes Mellitus in Obese; Cryotherapy Effect
Keywords: TII DM; Obese Females; Cryolipolysis
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryolipolysis Group (Active Comparator): About 30 obese females with type 2 diabetes and will face cryolypolysis in addition to exercise therapy treatment
  Interventions: Procedure: Cryolipolysis
- Group of Exercise (Active Comparator): About 30 obese females with type 2 diabetes and will face exercise therapy treatment only.
  Interventions: Procedure: Cryolipolysis

INTERVENTIONS:
Procedure: Cryolipolysis — To investigate the Effect of Cryolipolysis On insulin resistance and In adult type 2 female patients.
  Other Names: Exercise therapy

SUMMARY:
Diabetes mellitus (DM) is a complex chronic illness associated with a state of high blood glucose level, or hyperglycemia, occurring from deficiencies in insulin secretion, action, or both.

Diabetes mellitus is the name given to a wide spectrum group of disorders characterized by raised plasma glucose.Type 1 diabetes is characterized by an absolute insulin deficiency due to autoimmune destruction of insulin producing beta cells in the pancreas.

most adults with diabetes have type 2, characterized by a relative insulin secretory defect, and target tissue resistance to the effects of insulin.

DETAILED DESCRIPTION:
Diabetes is one of the most important health problems and chronic metabolic diseases requiring critical care.The number of people with diabetes has risen from 108 million in 1980 to 422 million in 2014.

Type 2 diabetes mellitus is a common and increasingly prevalent disease and is thus a major public health concern worldwide. The International Diabetes Federation estimates that there are approximately 387 million people diagnosed with diabetes across the globe.

The clinical diagnosis of diabetes is reliant on either one of the four plasma glucose (PG) criteria: elevated (i) fasting plasma glucose (FPG) (>126 mg/dL), (ii) 2 h PG during a 75-g oral glucose tolerance test (OGTT) (>200 mg/dL), (iii) random PG (>200 mg/dL) with classic signs and symptoms of hyperglycemia, or (iv) hemoglobin A1C level >6.5%.

The principal tissues affected by insulin resistance are liver, muscle and fat. In the liver this impaired insulin related inhibition of hepatic gluconeogenesis results in increased hepatic glucose output, exacerbating hyperglycemia.

In muscle, reduced transport of carbohydrates into muscle combined with lipid deposition in muscle cells leads toimpaired exercise ability and lowered threshold for tiredness with exercise. In fat tissue, there is impaired insulin-mediated inhibition of hormone dependent lipase, with breakdown of lipids to free fatty acids and glycerol, contributing to the dyslipidemia. With the rise in diabetes prevalence, researchers have increasingly investigated treatments intended to improve health and quality of life. People are much more likely to achieve metabolic control when they adhere to recommended diets, medications and exercise behaviors.

Cryolipolysis (CoolSculpting, Zeltiq, Pleasanton, CA) is a novel method of selective removal of fat with cooling. This technique is basedon the concept that fat cells are more sensitive to cold than the surrounding tissue. Prior studies and observations have demonstrated that cold exposure can induce selective damage to the subcutaneous fat via induction of panniculitis, resulting in reduction in the superficial fat layer of the skin

ELIGIBILITY:
Inclusion Criteria:

* Patients with incidence of diabetes 5 years ago.
* Patient fasting glucose level is more than 140 mg/dL.
* Age will be ranged from 35 to 45 years
* Body mass index between 25 and 30.
* All patients are medically controlled
* All patients have the same medical care.
* All patients will receive a good explanation of treatment procedures.

Exclusion Criteria:

* Patients dependent on insulin.
* Renal failure.
* Myocardial infractions.
* Cardiovascular problems.
* Neurological disorders.
* Patients with orthopedic problems (e.g mal or incomplete union of fracture, ankle sprains.
* Abdominal hernia
* Skin disease
* Unstable cases

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Skin fold thickness and estimation of total body fat | 3 months
  Estimation of body fat for all cases and is done by measuring these parameters :
  weight in kilograms, height in meters as weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Akram Abd El Aziz, Assist.Prof, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No